CLINICAL TRIAL: NCT04194177
Title: Evaluation of Two Types of Mechanical Ventilation During Robotic Surgery With the Thoracic Impedance Tomography
Brief Title: Evaluation of Thoracic Impedance Tomography During Robotic Surgery
Acronym: EIT_ROBO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Maria Vargas, resercher, Federico II University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: EIT_OR
Record Dates: First submitted 2019-12-08; First posted 2019-12-11 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Atelectasis
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- protective (Experimental)
  Interventions: Other: mechanical ventilation during robotic surgery
- conventional (Active Comparator)
  Interventions: Other: mechanical ventilation during robotic surgery

INTERVENTIONS:
Other: mechanical ventilation during robotic surgery — protective ventilation PEEP= 6 cmh2o TV= 6 ml/kg conventional PEEP=2 cmH2O and TV=9 ml/kg

SUMMARY:
the evaluation of distribution of mechanical ventilation during robotic surgery

ELIGIBILITY:
Inclusion Criteria:

* age>18
* informed consent
* robotic surgery

Exclusion Criteria:

* age<18
* no consent for the study

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
distribution of tidal volume | at the end of surgery

SECONDARY OUTCOMES:
driving pressure | at the end of surgery

CONTACTS AND LOCATIONS:
Locations (1):
- University of Naples Federico II department of Anesthesia and Critical Care, Naples, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Buonanno P, Marra A, Iacovazzo C, Merola R, De Siena AU, Servillo G, Vargas M. Electric impedance tomography and protective mechanical ventilation in elective robotic-assisted laparoscopy surgery with steep Trendelenburg position: a randomized controlled study. Sci Rep. 2023 Feb 16;13(1):2753. doi: 10.1038/s41598-023-29860-x. PMID 36797394